CLINICAL TRIAL: NCT02410902
Title: A Double Blind, Randomized, Placebo-Controlled Study of CM-AT for the Treatment of Autism in Children With All Levels of Fecal Chymotrypsin (FCT)
Brief Title: A Trial of CM-AT in Children With Autism With All Levels of FCT (The Blum Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Curemark (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00103
Record Dates: First submitted 2015-03-19; First posted 2015-04-08 (Estimated); Results first posted 2022-10-26 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2022-09

CONDITIONS: Autism
Keywords: Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CM-AT (Experimental): Active substance in single unit dose powder
  Interventions: Drug: CM-AT
- Placebo (Placebo Comparator): Placebo powder of inactive substance
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: CM-AT — Single unit dose powder of active substance (CM-AT) administered 3 times per day for 90 days
  Arms: CM-AT
Drug: PLACEBO — Single unit dose powder of non-active substance administered 3 times per day for 90 days
  Other Names: placebo powder
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether CM-AT is safe and effective in treating the core symptoms of autism in children with all levels of fecal chymotrypsin.

DETAILED DESCRIPTION:
Autism is clearly a significant cause of disability in the pediatric population. Many children with Autism exhibit impaired protein digestion which may or may not manifest in self-restricted diets. The inability to digest protein affects the availability of essential amino acids in the body. CM-AT is designed to enhance protein digestion thereby potentially restoring the pool of essential amino acids. Essential amino acids play a critical role in the expression of several genes important to neurological function and serve as precursors to key neurotransmitters such as serotonin and dopamine. CM-AT is a proprietary enzyme that is designed as a granulated powder taken three times daily.

ELIGIBILITY:
Inclusion Criteria:

* Meets the current Diagnostic and Statistical Manual with Mental Disorders (DSM-IV-TR) for Autism (Autistic Disorder), screened by SCQ and confirmed by ADI-R;

Exclusion Criteria:

* Patient weighing < 13kg (28.6 lbs)
* Previous allergy to porcine (pork) products
* Previous history of severe head trauma or stroke, loss of consciousness, seizure (or need for seizure medication either present or past) within one year of entering study or uncontrolled systemic disease
* Diagnosis of: HIV, cerebral palsy, endocrine disorder, pancreatic disease, muscular dystrophy, known genetic disorder, blood dyscrasia, ongoing GI disease
* Evidence of severe, moderate or uncontrolled systemic disease; and/or any co-morbid condition which in the Investigator's or Medical Director's opinion makes it undesirable for the subject to participate in the study or jeopardizes compliance with the protocol;
* Within 30 days of starting the study, certain supplementation, chelation or dietary restriction (a 30 day washout period would be required for inclusion);
* Ongoing dietary restriction for allergy or other reasons except nut allergies (lactose-free allowable);
* Use of of any stimulant medication must be discontinued 5 days prior to entering the study.
* Subject must have a stable dose of SSRI's for at least 30 days.
* Inability to ingest study drug and/or follow prescribed dosing schedule

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 190 (Actual)
Dates: Start 2015-05-13 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Pearson, PhD, Principal Investigator — The University of Texas Health Science Center, Houston; Robert Hendren, DO, Principal Investigator — University of California, San Francisco
Locations (31):
- United States (31):
  - Southwest Autism Research & Resource Center (S.A.R.R.C.), Phoenix, Arizona
  - University of Arizona, Pediatrics Multidisciplinary Research Unit, Tucson, Arizona
  - Arkansas Children'S Hosp. Research Institute (A.C.H.R.I.), Little Rock, Arkansas
  - N.R.C. Research Institute, Orange, California
  - M.I.N.D. Institute (Univ.of California, Davis), Sacramento, California
  - University of California (U.C.S.F.), San Francisco, California
  - IMMUNOe RESEARCH CENTERS, Centennial, Colorado
  - Yale Child Study Center, New Haven, Connecticut
  - Segal Institute For Clinical Research, North Miami, Florida
  - Florida Hospital Medical Group-Lake Mary Pediatrics, Orange City, Florida
  - Kaley Kildahl, Orlando, Florida
  - Research Institute of Deaconess Clinic, Evansville, Indiana
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - L.S.U. Health Sciences Center, Shreveport, Louisiana
  - Detroit Clinical Research Center, P.C., Bingham Farms, Michigan
  - Children'S Specialized Hospital, Egg Harbor, New Jersey
  - Children'S Specialized Hospital, Toms River, New Jersey
  - Clinical Research Center of Nj, Voorhees Township, New Jersey
  - Lovelace Scientific Resources, Albuquerque, New Mexico
  - Richmond Behavioral Associates, Staten Island, New York
  - Montefiore Med.Center, Autism & Obsessive Compulsive Spectrum Prog., The Bronx, New York
  - Duke Center For Autism and Brain Development, Durham, North Carolina
  - Cleveland Clinic, Center For Autism Research, Cleveland, Ohio
  - Omega Medical Research, Warwick, Rhode Island
  - Carolina Clinical Trials, Inc., Charleston, South Carolina
  - Vanderbilt University Med.Center -Treatment & Research Inst. For Asd, Nashville, Tennessee
  - University of Texas, Houston Dept. of Psychiatry and Behavioral Sciences, Houston, Texas
  - Ericksen Research & Development, Clinton, Utah
  - University of Virginia, Dept. of Psychiatry and Neurobehavioral Sciences, Charlottesville, Virginia
  - Neuroscience, Inc., Herndon, Virginia
  - Carilion Clinic-Virginia Tech, Carilion School of Medicine, Roanoke, Virginia

REFERENCES:
- [Background] McPheeters ML, Warren Z, Sathe N, Bruzek JL, Krishnaswami S, Jerome RN, Veenstra-Vanderweele J. A systematic review of medical treatments for children with autism spectrum disorders. Pediatrics. 2011 May;127(5):e1312-21. doi: 10.1542/peds.2011-0427. Epub 2011 Apr 4. PMID 21464191
- [Background] Autism and Developmental Disabilities Monitoring Network Surveillance Year 2008 Principal Investigators; Centers for Disease Control and Prevention. Prevalence of autism spectrum disorders--Autism and Developmental Disabilities Monitoring Network, 14 sites, United States, 2008. MMWR Surveill Summ. 2012 Mar 30;61(3):1-19. PMID 22456193
- [Background] Developmental Disabilities Monitoring Network Surveillance Year 2010 Principal Investigators; Centers for Disease Control and Prevention (CDC). Prevalence of autism spectrum disorder among children aged 8 years - autism and developmental disabilities monitoring network, 11 sites, United States, 2010. MMWR Surveill Summ. 2014 Mar 28;63(2):1-21. PMID 24670961
- [Background] Peacock G, Amendah D, Ouyang L, Grosse SD. Autism spectrum disorders and health care expenditures: the effects of co-occurring conditions. J Dev Behav Pediatr. 2012 Jan;33(1):2-8. doi: 10.1097/DBP.0b013e31823969de. PMID 22157409
- [Background] Ganz ML. The lifetime distribution of the incremental societal costs of autism. Arch Pediatr Adolesc Med. 2007 Apr;161(4):343-9. doi: 10.1001/archpedi.161.4.343. PMID 17404130
- [Background] McElhanon BO, McCracken C, Karpen S, Sharp WG. Gastrointestinal symptoms in autism spectrum disorder: a meta-analysis. Pediatrics. 2014 May;133(5):872-83. doi: 10.1542/peds.2013-3995. PMID 24777214
- [Background] Buie T, Campbell DB, Fuchs GJ 3rd, Furuta GT, Levy J, Vandewater J, Whitaker AH, Atkins D, Bauman ML, Beaudet AL, Carr EG, Gershon MD, Hyman SL, Jirapinyo P, Jyonouchi H, Kooros K, Kushak R, Levitt P, Levy SE, Lewis JD, Murray KF, Natowicz MR, Sabra A, Wershil BK, Weston SC, Zeltzer L, Winter H. Evaluation, diagnosis, and treatment of gastrointestinal disorders in individuals with ASDs: a consensus report. Pediatrics. 2010 Jan;125 Suppl 1:S1-18. doi: 10.1542/peds.2009-1878C. PMID 20048083
- [Background] Samsam M, Ahangari R, Naser SA. Pathophysiology of autism spectrum disorders: revisiting gastrointestinal involvement and immune imbalance. World J Gastroenterol. 2014 Aug 7;20(29):9942-51. doi: 10.3748/wjg.v20.i29.9942. PMID 25110424
- [Background] Elsabbagh M, Divan G, Koh YJ, Kim YS, Kauchali S, Marcin C, Montiel-Nava C, Patel V, Paula CS, Wang C, Yasamy MT, Fombonne E. Global prevalence of autism and other pervasive developmental disorders. Autism Res. 2012 Jun;5(3):160-79. doi: 10.1002/aur.239. Epub 2012 Apr 11. PMID 22495912
- [Background] Wasfy M, Oyofo B, Elgindy A, Churilla A. Comparison of preservation media for storage of stool samples. J Clin Microbiol. 1995 Aug;33(8):2176-8. doi: 10.1128/jcm.33.8.2176-2178.1995. PMID 7559972
- [Background] Cavallini G, Benini L, Brocco G, Riela A, Bovo P, Pederzoli P, Angelini G, Pelle C, Bertelli G, Scuro LA. The fecal chymotrypsin photometric assay in the evaluation of exocrine pancreatic capacity. Comparison with other direct and indirect pancreatic function tests. Pancreas. 1989;4(3):300-4. doi: 10.1097/00006676-198906000-00005. PMID 2734275
- [Background] Matthews DM. Intestinal absorption of amino acids and peptides. Proc Nutr Soc. 1972 Sep;31(2):171-7. doi: 10.1079/pns19720033. No abstract available. PMID 4563292
- [Background] Coutinho AM, Oliveira G, Morgadinho T, Fesel C, Macedo TR, Bento C, Marques C, Ataide A, Miguel T, Borges L, Vicente AM. Variants of the serotonin transporter gene (SLC6A4) significantly contribute to hyperserotonemia in autism. Mol Psychiatry. 2004 Mar;9(3):264-71. doi: 10.1038/sj.mp.4001409. PMID 15094787
- [Background] Naushad SM, Jain JM, Prasad CK, Naik U, Akella RR. Autistic children exhibit distinct plasma amino acid profile. Indian J Biochem Biophys. 2013 Oct;50(5):474-8. PMID 24772971
- [Background] Tang G, Gudsnuk K, Kuo SH, Cotrina ML, Rosoklija G, Sosunov A, Sonders MS, Kanter E, Castagna C, Yamamoto A, Yue Z, Arancio O, Peterson BS, Champagne F, Dwork AJ, Goldman J, Sulzer D. Loss of mTOR-dependent macroautophagy causes autistic-like synaptic pruning deficits. Neuron. 2014 Sep 3;83(5):1131-43. doi: 10.1016/j.neuron.2014.07.040. Epub 2014 Aug 21. PMID 25155956
- [Background] Balasubramanian MN, Butterworth EA, Kilberg MS. Asparagine synthetase: regulation by cell stress and involvement in tumor biology. Am J Physiol Endocrinol Metab. 2013 Apr 15;304(8):E789-99. doi: 10.1152/ajpendo.00015.2013. Epub 2013 Feb 12. PMID 23403946
- [Background] Fairclough PD, Hegarty JE, Silk DB, Clark ML. Comparison of the absorption of two protein hydrolysates and their effects on water and electrolyte movements in the human jejunum. Gut. 1980 Oct;21(10):829-34. doi: 10.1136/gut.21.10.829. PMID 7192244
- [Background] Arnold GL, Hyman SL, Mooney RA, Kirby RS. Plasma amino acids profiles in children with autism: potential risk of nutritional deficiencies. J Autism Dev Disord. 2003 Aug;33(4):449-54. doi: 10.1023/a:1025071014191. PMID 12959424
- [Background] Munasinghe SA, Oliff C, Finn J, Wray JA. Digestive enzyme supplementation for autism spectrum disorders: a double-blind randomized controlled trial. J Autism Dev Disord. 2010 Sep;40(9):1131-8. doi: 10.1007/s10803-010-0974-2. PMID 20204691
- [Background] Schreck KA, Williams K, Smith AF. A comparison of eating behaviors between children with and without autism. J Autism Dev Disord. 2004 Aug;34(4):433-8. doi: 10.1023/b:jadd.0000037419.78531.86. PMID 15449518
- [Background] Bailey DB Jr, Raspa M, Olmsted M, Holiday DB. Co-occurring conditions associated with FMR1 gene variations: findings from a national parent survey. Am J Med Genet A. 2008 Aug 15;146A(16):2060-9. doi: 10.1002/ajmg.a.32439. PMID 18570292
- [Background] Lecavalier L. An evaluation of the Gilliam Autism Rating Scale. J Autism Dev Disord. 2005 Dec;35(6):795-805. doi: 10.1007/s10803-005-0025-6. PMID 16283084
- [Background] Marcus RN, Owen R, Kamen L, Manos G, McQuade RD, Carson WH, Aman MG. A placebo-controlled, fixed-dose study of aripiprazole in children and adolescents with irritability associated with autistic disorder. J Am Acad Child Adolesc Psychiatry. 2009 Nov;48(11):1110-1119. doi: 10.1097/CHI.0b013e3181b76658. PMID 19797985
- [Background] Yerys BE, Wallace GL, Sokoloff JL, Shook DA, James JD, Kenworthy L. Attention deficit/hyperactivity disorder symptoms moderate cognition and behavior in children with autism spectrum disorders. Autism Res. 2009 Dec;2(6):322-33. doi: 10.1002/aur.103. PMID 19998356
- [Background] Schreck KA, Williams K. Food preferences and factors influencing food selectivity for children with autism spectrum disorders. Res Dev Disabil. 2006 Jul-Aug;27(4):353-63. doi: 10.1016/j.ridd.2005.03.005. Epub 2005 Jul 25. PMID 16043324
- [Background] Borowitz D. Update on the evaluation of pancreatic exocrine status in cystic fibrosis. Curr Opin Pulm Med. 2005 Nov;11(6):524-7. doi: 10.1097/01.mcp.0000181474.08058.b3. PMID 16217179
- [Background] Penn AH, Hugli TE, Schmid-Schonbein GW. Pancreatic enzymes generate cytotoxic mediators in the intestine. Shock. 2007 Mar;27(3):296-304. doi: 10.1097/01.shk.0000235139.20775.7f. PMID 17304111
- [Background] Williams K, Wheeler DM, Silove N, Hazell P. Selective serotonin reuptake inhibitors (SSRIs) for autism spectrum disorders (ASD). Cochrane Database Syst Rev. 2010 Aug 4;(8):CD004677. doi: 10.1002/14651858.CD004677.pub2. PMID 20687077
- [Derived] Pearson DA, Hendren RL, Heil MF, McIntyre WR, Raines SR. Pancreatic Replacement Therapy for Maladaptive Behaviors in Preschool Children With Autism Spectrum Disorder. JAMA Netw Open. 2023 Nov 1;6(11):e2344136. doi: 10.1001/jamanetworkopen.2023.44136. PMID 38032645

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited across 33 sites in the USA. The First Subject First Visit (FSFV) occurred on 03 June 2015 (First screening visit date) and the Last Subject Last Visit (LSLV) occurred on 20 December 2017.
Pre-assignment Details: Participants were screened for autistic disorder using the Diagnostic Statistical Manual of Mental Disorders Fourth Edition - Text Revised (DSM-IV-TR); and the Social Communication Questionnaire (SCQ), with diagnostic confirmation by the Autism Diagnostic Interview-Revised (ADI-R). All qualifying participants were given a 2 week run-in period and then reassessed for eligibility and then randomized.
Groups:
- CM-AT: Active substance in single unit dose powder
  CM-AT: Single unit dose powder of active substance, 900mg, (CM-AT) administered 3 times per day, one at each meal for 90 days. Participants were between 3 and 8 years old inclusive.
- Placebo: Placebo powder of inactive substance
  PLACEBO: Single unit dose powder of non-active substance, 900mg, (Placebo) administered 3 times per day, one at each meal for 90 days. Participants were between 3 and 8 years old inclusive.
Period: Overall Study
Arm/Group | CM-AT | Placebo
Started | 92 | 98
Randomized | 92 | 98
ITT | 92 | 98
Completed | 71 | 80
Not Completed | 21 | 18
Not completed — Adverse Event | 2 | 3
Not completed — Lost to Follow-up | 4 | 1
Not completed — Protocol Violation | 1 | 4
Not completed — Withdrawal by Subject | 6 | 8
Not completed — Non-Compliance | 8 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CM-AT | Placebo | Total
Number analyzed (Participants) | 92 | 98 | 190
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 92 | 98 | 190
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 5.7 (1.6) | 5.7 (1.6) | 5.7 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 40
  Male | 71 | 79 | 150
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 80 | 100
  Not Hispanic or Latino | 71 | 18 | 89
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 12 | 10 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 8 | 18
  White | 61 | 70 | 131
  More than one race | 7 | 6 | 13
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 92 | 98 | 190
ABC-I [Mean (Standard Deviation); unit: units on a scale] — The ABC-I is a discrete sub scale of the Aberrant Behavior Checklist (ABC) - Community. The "I" is the Irritability sub scale. Scale range is 0-45. A higher score reflects higher severity of symptoms (irritability). The Baseline measurement indicates the subject's initial score on this sub scale. Scores are obtained via Parent Rated Questionnaire. Parents respond to a series of questions on scale (0 = not at all a problem 1 = the behavior is a problem but slight in degree 2 = the problem is moderately serious 3 = the problem is severe in degree). Questions correspond to one of 5 sub scales.
  units on a scale | 22.2 (7.6) | 23.4 (7.9) | 22.8 (7.75)

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome Measurements to Determine Efficacy of Treatment With CM-AT Versus Placebo for Changes in the Aberrant Behavior Checklist Subscale for Irritability / Agitation (ABC-I) Between Baseline and Week 12/Termination Visit
Description: Primary outcome measurements to determine efficacy of treatment with CM-AT versus Placebo for changes in the Aberrant Behavior Checklist (ABC) - Community sub scale for Irritability/Agitation (ABC-I) between baseline (subject's initial measurement) and Week 12/Termination (subject's final measurement) visit. Participants were between 3 through to 6 years old inclusive and took 900mg CM-AT or Placebo three times daily. The ABC-I is one of five discrete sub scales measured by the ABC. The scale range is 0-45. A higher score reflects higher severity of symptoms (irritability). Scores are obtained via Parent Rated Questionnaire. Parents respond to a series of questions on a scale directly into an electronic data capture system (EDC), responding: 0 = not at all a problem 1 = the behavior is a problem but slight in degree 2 = the problem is moderately serious 3 = the problem is severe in degree. The score was automatically calculated by the EDC.
Time Frame: Screening through Week 12/Termination
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- CM-AT: Active substance in single unit dose powder
  Participants were between 3 through to 6 years old inclusive and took 900mg CM-AT. Participants took 3 sachets of CM-AT in total: One at each meal
- Placebo: Placebo powder of inactive substance
  Participants were between 3 through to 6 years old inclusive and took 900mg Placebo. Participants took 3 sachets of Placebo in total: One at each meal
Arm/Group | CM-AT | Placebo
Number analyzed (Participants) | 92 | 98
units on a scale | -8.0 (7.47) | -5.5 (9.19)
Statistical Analysis 1: Comparison: CM-AT vs Placebo; Test type: Other — ANCOVA using MMRM analysis; p = 0.038, ANCOVA; Mean Difference (Final Values) = -2.56, 95% CI 2-sided [-4.98 to -0.14]

2. Secondary Outcome: Secondary Outcome Measurements of Changes in the Aberrant Behavior Checklist Checklist Subscale for Lethargy / Social Withdrawal (ABC-L) Between Baseline and Week 12/Termination Visit
Description: Secondary outcome measurements to determine efficacy of treatment with CM-AT versus Placebo for changes in the Aberrant Behavior Checklist- Community (ABC) sub scale for Lethargy / Social Withdrawal (ABC-L) between baseline (subject's initial measurement) and Week 12/Termination (subject's final measurement) visit. Participants were between 3 through to 6 years old inclusive and took 900mg CM-AT or Placebo three times daily. The ABC-L is one of five discrete sub scales measured by the ABC. The scale range is 0-48. A higher score reflects higher severity of symptoms (lethargy). Scores are obtained via Parent Rated Questionnaire. Parents respond to a series of questions on a scale directly into an electronic data capture system (EDC), responding: 0 = not at all a problem 1 = the behavior is a problem but slight in degree 2 = the problem is moderately serious 3 = the problem is severe in degree.
Time Frame: Screening through Week 12/Termination.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CM-AT | Placebo
Number analyzed (Participants) | 92 | 98
units on a scale | -7.9 (6.96) | -6.6 (9.52)
Statistical Analysis 1: Comparison: CM-AT vs Placebo; Test type: Other — ANCOVA using MMRM analysis; p = 0.325, ANCOVA; Mean Difference (Final Values) = -1.07, 95% CI 2-sided [-3.21 to 1.07]

ADVERSE EVENTS:
Time Frame: Adverse Events were recorded from the time of consent through 30-days following subject completion of or withdrawal from study, equalling a maximum of 128 days.
Arm/Group | CM-AT | Placebo
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/98
Serious Adverse Events (participants affected / at risk) | 0/92 | 0/98
Other Adverse Events (participants affected / at risk) | 79/92 | 90/98
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CM-AT (N=92) | Placebo (N=98)
Nasopharyngitis (Infections and infestations) | 24 (28) | 28 (35)
Stool pH Decreased (Investigations) | 15 (17) | 22 (28)
Constipation (Gastrointestinal disorders) | 17 (25) | 14 (18)
Pyrexia (General disorders) | 15 (22) | 17 (27)
Vomiting (Gastrointestinal disorders) | 11 (12) | 14 (16)
Diarrhoea (Gastrointestinal disorders) | 5 (10) | 14 (17)
Upper Respiratory Tract Infections (Infections and infestations) | 11 (16) | 14 (19)
Stool Analysis Abnormal (Investigations) | 3 | 11
Clostridium Test Positive (Investigations) | 7 (8) | 8 (8)
Headache (Nervous system disorders) | 4 (5) | 5 (7)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 10 (13) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 8 (12)
Stool pH Increased (Investigations) | 4 (4) | 12
Ear Pain (Ear and labyrinth disorders) | 8 (8) | 1
Seasonal Allergy (Immune system disorders) | 5 (5) | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications include input from PI and Curemark reflected in authorship. Institution's results may be submitted after results of the multicenter study are published, 18m after completion, or if multicenter publication isn't planned. Then PI may to publish, subject to confidentiality agreement. PI shall give to Curemark 45 days prior for review. Submission of such publication of results be can't delayed more than 105d after being received by Curemark. After 105 days, the PI may publish.

DOCUMENTS (2):
  • Study Protocol (2017-02-17): https://cdn.clinicaltrials.gov/large-docs/02/NCT02410902/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-27): https://cdn.clinicaltrials.gov/large-docs/02/NCT02410902/SAP_001.pdf